CLINICAL TRIAL: NCT03523611
Title: Cardiac Magnetic Resonance Assessment of Right Ventricular Inflammation After Lung Resection - a Feasibility Study
Brief Title: Right Ventricular Inflammation After Lung Resection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Dr Ben Shelley, Consultant Cardio-thoracic Anaesthesia and Critical Care, University of Glasgow
Other Study IDs: 17/ANAES/06
Record Dates: First submitted 2018-04-18; First posted 2018-05-14 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Lung Cancer; Ventricular Failure
Keywords: lung cancer; Ventricular Failure
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- lung resection: Patients with suspected lung cancer undergoing lung resection by anatomic lobectomy
  Interventions: Procedure: Lung Resection

INTERVENTIONS:
Procedure: Lung Resection — Lung resection surgery

SUMMARY:
The purpose of this study is explore the impact of lung cancer surgery on inflammation and function of the right side of the heart.

DETAILED DESCRIPTION:
Lung cancer is the second most common cancer in the UK and is the leading cause of cancer related death. Where appropriate, surgery to remove the tumour and the surrounding lung (lung resection) provides the best chance of cure. Frequently patients are either current or ex-smokers with related lung or heart problems which increase the risks associated with surgery. Following surgery patients may suffer long term shortness of breath, greatly limiting their day-to-day function and lowering quality of life. The investigators believe this shortness of breath is not solely caused by the removal of part of the lung but also from a decrease in the performance of the heart. Although the surgery does not directly involve the heart it is thought that the damage is caused indirectly by the surgery and by the removal of part of the lung.

In a previous study, the investigators showed that the function of the right side of the heart (the right heart) is decreased following lung resection. The decrease in right heart (the part that supplies blood to the lungs) function was associated with a prolonged stay in the high dependency unit and blood markers indicating damage to the heart. The process by which the damage occurs is poorly understood, but it is thought that an increase in the forces preventing the right heart pumping blood (resistance) is to blame. The decrease in function in the right heart may be triggered during surgery by the diminished blood supply to the cancerous lung and, and maintained post operatively, as lung resection can cause a long-term increase in resistance.

Diseases that cause an increase in resistance to the right heart have been shown to cause damage to different parts of the right heart. An acute sudden increase in resistance can cause inflammation, thinning and scarring whilst a long-term increase in resistance causes the right heart to thicken. The investigators believe that the potential damage during the operation could cause permanent damage to the right heart and contribute to shortness of breath and functional limitation.

To investigate the potential inflammation/scarring and the function of the heart the investigators will image the heart with specialised Magnetic Resonance Imaging (MRI) scans.

The aim of the research is to determine whether inflammation occurs in the right heart during and following lung resection and, if so, does it result in scarring?. The investigators will compare the function of the right heart before, during and after surgery to determine if inflammation contributes to the decrease in right heart function following lung resection seen in our previous study. The investigators anticipate that the study will increase understanding of how the right heart may be damaged by lung resection. The investigators believe this will guide further studies aiming to prevent such damage, ultimately limiting the disabling breathlessness and decrease in heart function that so greatly affects patients' lives.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent
2. Age >16 years
3. Planned elective lung resection by VATS or open lobectomy

Exclusion Criteria:

1. Pregnancy
2. On-going participation in any investigational research which could undermine the scientific basis of the study
3. Wedge, segmental or sub-lobar lung resection
4. Pneumonectomy
5. Isolated right middle lobectomy
6. Atrial fibrillation at baseline
7. Contraindication to cardiac magnetic resonance imaging

   1. Cardiac pacemaker, artificial heart valve, neurostimulator, cochlear implant
   2. Aneurysm clips
   3. Metal injuries to the eye
   4. Loose metal in a part of the body
8. Contraindication to IV Gadolinium (contrast) administration:

   1. Acute or chronic renal failure
   2. Allergy to contrast

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing lobectomy for primary lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2018-04-30 (Actual); Primary Completion 2019-04-19 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Can RV inflammation be assessed by T1 mapping CMR following lung resection by assessing the number of CMR studies which have an IQS>1? | 2 months
  The investigators will test and report inter- and intra-observer reproducibility of Region of Interest (ROI) definition in all datasets where Image Quality Score (IQS)>1. The primary endpoint will be the number of MRI studies which have an IQS >1.

SECONDARY OUTCOMES:
Are T1 values at the ventricular insertion points increased following lung resection? | 2 months
  In all patients, the investigators willl measure T1 values at the ventricular insertion points using ROI tool to determine if T1 is increased following lung resection.
Association between RV inflammation and RV fibrosis following lung resection using measurement of extracellular volume? | 2 months
  Does the presence of RV inflammation ultimately lead to the development of RV fibrosis. In all patients, ECV will be assessed. An increase in ECV indicates development of fibrosis
Is there any evidence of inflammation/fibrosis in the LV? | 2 months
  T1 values will be assessed in all patients at the LV free wall using ROI tool. ECV at the LV free wall will be measured to determine if there is fibrosis present.

CONTACTS AND LOCATIONS:
Locations (1):
- Golden Jubilee National Hospital, Glasgow, Strathclyde, United Kingdom

IPD SHARING:
Plan to Share IPD: No